CLINICAL TRIAL: NCT06853314
Title: An Effectiveness Trial of WINGS+PrEP: a Syndemic mHealth Intervention to Increase PrEP Uptake Among Women Impacted by Heavy Alcohol Use and Partner Violence in the Criminal Legal System
Brief Title: An Effectiveness Trial of the PrEP for WINGS Study
Acronym: PFW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anindita Dasgupta, Assistant Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU7312; 1R01AA030462 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Alcohol Use Disorder; Violence, Gender-Based
Keywords: Intimate partner violence; Hazardous alcohol use; HIV infection; PrEP
MeSH Terms: conditions — HIV Infections; Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEP for WINGS (intervention arm) (Experimental): Participants randomized to the PrEP for WINGS intervention arm will receive three sessions on a self-paced intervention delivered via a mobile health platform. Session 1 will focus on HIV risk reduction and deliver the PrEP Decision Aid. Sessions 2-3 will involve sessions focused on IPV and alcohol SBIRT sessions with peer navigation that will be completed within a 30 day period (3 sessions total). PrEP for WINGS mHealth sessions may be delivered using smart phones or using tablets available at study data collection sites. Intervention participants will also receive three peer navigation sessions from Community Health Advocates who will help participants trouble shoot any barriers to linking to care, and meeting goals set during the intervention sessions.
  Interventions: Behavioral: PrEP for WINGS
- PrEP alone (control arm) (Active Comparator): Participants randomized to the control arm of the study will receive a single session on HIV risk reduction and the patient-centered PrEP Decision Aid. This individual session will be identical to the first session of the PrEP for WINGS three session intervention, and will also be delivered through an online survey platform. In addition, study participants in the control condition will also have one peer navigation session with a Community Health Advocate at the end of the self-paced session to help facilitate linkage to care.
  Interventions: Behavioral: PrEP Decision Aid

INTERVENTIONS:
Behavioral: PrEP for WINGS — The PrEP for WINGS intervention involves three sessions of a self-paced and self-directed intervention delivered via a mobile health platform. Session 1 will focus on HIV risk reduction and provide the PrEP Decision Aid, where participants will learn information about PrEP to help them decide if it is appropriate for them. Sessions 2-3 will involve integrated Screening, Brief Intervention, Referral to Treatment (SBIRT) modules focused on IPV and alcohol reduction. The PrEP for WINGS intervention will also involve peer navigation sessions with Community Health Advocates to help intervention participants trouble shoot any barriers to achieving goals they set during the self-paced sessions. The PrEP for WINGS intervention will take place over a 30 day period and Sessions 2-3, and the peer navigation sessions may be delivered using smart phones or using tablets available at study data collection sites.
  Arms: PrEP for WINGS (intervention arm)
Behavioral: PrEP Decision Aid — The PrEP Decision Aid will be delivered to participants in the control condition, and focus on helping study participants decide if they should initiate PrEP. This single session will focus on HIV risk reduction, and then launch the patient-centered PrEP Decision Aid. This individual session will be identical to the first session of the PrEP for WINGS three session intervention, and will also be delivered through an online survey platform. In addition, study participants in the control condition will also have one peer navigation session with a Community Health Advocate at the end of the self-paced session to help facilitate linkage to care.
  Arms: PrEP alone (control arm)

SUMMARY:
(Effectiveness Aim 1) To test the comparative effectiveness of PreP for WINGS versus PrEP alone on primary outcomes of increasing PrEP initiation measured by self-report/medical records, recent adherence measured by urine assay of Tenofovir (TDF) and longer-term adherence by self-report/medical records over the 12-month follow-up; and secondary outcomes of decreasing IPV, hazardous drinking, recidivism, and HIV risks.

(Moderation Aim 2) To test if the effectiveness of WINGS+PrEP on study outcomes is moderated by key participant subgroups based on race/ethnicity, sexual orientation, age, education, incarceration history, IPV severity, substance use disorders (SUDs), digital access and literacy, housing stability, and medical mistrust.

DETAILED DESCRIPTION:
This hybrid type 1 Effectiveness and Implementation Trial will evaluate an m-Health syndemic intervention (PrEP for WINGS) that aims to increase HIV pre-exposure prophylaxis (PrEP) initiation and adherence among women in community supervision programs (CSPs) including probation, parole, and alternative-to-incarceration (ATI) programs) in New York City (NYC) who report hazardous drinking. PrEP is a proven effective biomedical strategy to prevent HIV infection. To date, however, very few PrEP interventions have focused on cis-gender women, and none have targeted women in CSPs, who due to racialized drug laws, are disproportionately Black and Latinx. Women in CSPs have high rates of HIV risk behaviors (e.g., frequent condomless sex, sex with multiple partners) and elevated rates of HIV infection as high as 17%. Large racial health disparities in PrEP uptake exist, a nationally representative study showing that Black women in the USA were four times less likely to have initiated PrEP than non-Hispanic white women. Advancing an effective PrEP intervention for women in CSPs holds promise for reducing HIV disparities by reaching a large number of Black and Latinx women who remain at high risk for HIV.

Compared to the general population, women in CSPs have very high rates of co-occurring hazardous drinking and intimate partner violence (IPV), which are major syndemic drivers of HIV infection and well-established barriers to PrEP uptake. PrEP enables women to engage in a female-controlled HIV prevention strategy, which is vitally important within the context of hazardous drinking and violent partners. To date, however, there are no evidence-based syndemic-focused PrEP interventions for women that address hazardous drinking and IPV exposure. The PrEP for WINGS intervention is a 3-session syndemic-focused intervention that combines an evidence-based mHealth Alcohol Screening, Brief Intervention, and Referral to Treatment (SBIRT) tool, and an evidence-based mHealth IPV SBIRT tool - WINGS (Women Initiating New Goals of Safety) with an evidence-based PrEP intervention that includes a PrEP decision making aid with novel PrEP telemedicine and peer navigation components delivered by Community Health Advocates (CHA). Peer navigation has been shown to increase PrEP initiation and adherence and reduce barriers related to medical mistrust and stigma, which is important for Black and Latinx women. The same single session evidence-based PrEP intervention with peer navigation will serve as the comparison condition (PrEP alone), allowing us to compare the added value of the WINGS syndemic components and offering a cost-efficient alternative evidence-based PrEP intervention. Both interventions will be implemented at various community-based organizations supporting women in CSPs in NYC.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a cis-gender woman
* Aged 18 or older
* Test negative for HIV using a rapid OraSure oral test at screening
* Are currently on probation, parole or an ATI programs as verified by CSP records
* Score positive for risk of hazardous drinking or alcohol dependence on AUDIT with a cut off score of 6 or higher; or indicated they drank 4 or more drinks on one occasion in the past 30 days
* Report ever experiencing any intimate partner violence (HARK score of ≤1)
* Report not taking PrEP in the past 90 days
* Report having had condomless vaginal or anal sex in the past 90 days; and report an outside HIV risk in the past year (i.e. sex with more than one partner, shared injected equipment, tested positive for a bacterial STI, had sex with a man with HIV and not virally suppressed).

Exclusion Criteria:

* Ability to speak and understand English is not sufficient to participate in assessments or intervention sessions.
* Inability to complete informed consent process due to a psychiatric or cognitive impairment (assessed by the Mini Folstein exam)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of completed PrEP provider meetings (PrEP Initiation) | From enrollment (baseline) to the end of 12-month follow up
  Meeting with a PrEP provider to start PrEP once will meet the threshold for PrEP initiation.

SECONDARY OUTCOMES:
Revised Conflict Tactic Scale Score | From enrollment (baseline) to the end of 12-month follow up
  This is designed to assess intimate partner violence (IPV) based on self-reporting on quantitative behavioral survey assessments using the Revised Conflict Tactic Scale 2. Questions are asked for 21 behaviors occurring in the three time frames prior to assessment: ever, past year, and past six months. Positive endorsement of any item will be scored with 1; negative endorsements will be scored 0. Scores range from 0 to 21 for each timeframe, with low score indicated fewer episodes of IPV in the given timeframe, where higher scores indicate higher number of episodes of IPV.
AUDIT Score | From enrollment (baseline) to the end of 12-month follow up
  The self-report version of the AUDIT will be used to assess hazardous alcohol use. The AUDIT has 10 questions and the possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Anindita Dasgupta, MPH, PhD, Principal Investigator — Columbia University; Louisa Gilbert, MSW, PhD, Principal Investigator — Columbia University; Rachel Groth, MSW, MPH, Study Director — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided